CLINICAL TRIAL: NCT04077346
Title: Neuromodulation of Spinal Locomotor Circuitry to Elicit Stepping After Pediatric Spinal Cord Injury
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Kentucky Spinal Cord and Head Injury Research Trust and Board (Unknown); Kosair Charities, Inc. (Other)
Responsible Party: Principal Investigator, Andrea L. Behrman, PhD, PT, Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19.0844
Record Dates: First submitted 2019-08-21; First posted 2019-09-04 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries
Keywords: Pediatric-onset; Transcutaneous spinal stimulation; Stepping
MeSH Terms: conditions — Spinal Cord Injuries; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Transcutaneous Spinal Stimulation- Acute and with Training. (Experimental): For Aim 1: Participants will receive transcutaneous stimulation (TcStim) in supine or side lying position at a single or multi site spinal levels to produce stepping/locomotor activity in lower limbs.
  For Aim 2: TcStim will be delivered while participants are stepping on a computerized treadmill with an overhead partial body weight support (BWS) system and while stepping overground.
  For Aim 3: Participants will first receive a combination of Activity-based locomotor training (AB-LT)+TcStim for 60 sessions.
  Interventions: Device: Biostim-5 transcutaneous spinal stimulator; Other: Transcutaneous Spinal Stimulator + Activity Based Locomotor Training

INTERVENTIONS:
Device: Biostim-5 transcutaneous spinal stimulator — Transcutaneous spinal stimulation (TcStim): The 5-channel stimulator capable of generating (41) pain-free biphasic rectangular waveform of 0.3- to 1.0-ms pulses with a frequency of 5-10 kHz will be used to stimulate at single or multi-site spinal levels.
  TcStim will be delivered in combination with activity based locomotor training in 5 - 10 minute of stimulation at sub-motor threshold daily (5x/week) for 60 sessions
Other: Transcutaneous Spinal Stimulator + Activity Based Locomotor Training — Participants will receive a combination of Activity-based locomotor training (AB-LT)+TcStim daily (5x/week) for 60 sessions and will consist of a minimum of 55-60 min on the TM for facilitated standing/stepping followed by 30 min of activities off TM in sitting, standing, or stepping.

SUMMARY:
Spinal cord injury (SCI) results in damage to the descending neural pathways and leads to the immediate dysfunction of multiple physiological systems below the level of injury. Like adults, children with SCI suffer from neuromuscular paralysis which results in the inability to sit, stand, and walk. Current therapeutic interventions largely aim to compensate for paralysis to achieve mobility based on the assumption that damage to the central nervous system is permanent and irreversible, e.g. use of braces, standers, and wheelchairs. The objective of this proposal is to investigate the use of transcutaneous spinal stimulation (TcStim) to enable stepping in children with chronic SCI.

The investigators will recruit 8 participants, ages 4-12 years with chronic, acquired SCI, T10 and above and non-ambulatory. The aims of this proposal are to 1) investigate the mechanisms of locomotor-specific regulation in the spinal neural circuitry of children with acquired SCI using single vs. multi-site TcStim, 2) investigate the capacity of the lumbosacral spinal cord for integration of task-specific input (e.g. load, speed) during facilitated stepping with and without TcStim, and 3) investigate the training effects of TcStim on the ability to step. Outcomes will provide a necessary initial step in the translation of scientific findings for neuromodulation from adults with SCI to children.

DETAILED DESCRIPTION:
Like in adults, children with spinal cord injury (SCI) in children suffer from neuromuscular paralysis which results in the inability to sit, stand, and walk. Current therapeutic interventions, e.g. leg braces, wheelchairs, largely aim to compensate for paralysis based on the assumption that damage to the central nervous system is permanent and irreversible.The discovery of the "intelligent" spinal cord, known as the central pattern generator (CPG), has demonstrated that complex neuronal networks are capable of generating rhythmic and coordinated motor patterns and has set forth a major paradigm shift in the investigators expectation of the possibility for recovery even with severe SCI. Studies have demonstrated, first, that after SCI, the CPG can be "accessed", reactivated, and retrained via sensory feedback arising from the muscles and joints during activity-based locomotor training (AB-LT). Second, application of epidural and transcutaneous stimulation (TcStim) to the spinal cord below the level of lesion can augment the neuromuscular capacity for voluntary movement, standing and stepping in adults with chronic motor complete SCI. While neural mechanisms for stepping regulation have been demonstrated in adults testing single vs. multi-site stimulation, this inherent capacity must be examined in children with SCI. Similarly, the addition of stimulation during AB-LT in adults with motor complete SCI has resulted in remarkable recovery of over ground walking. The immediate and long-term response of such combined therapeutic exposure and subsequent training has yet to be examined in children. Children with SCI may not only benefit from these novel therapeutic approaches but also demonstrate greater improvements in neuromuscular recovery due to inherent plasticity. The investigators' preliminary work has demonstrated the safety and feasibility of TcStim in children with SCI. Therefore, the specific aims of this proposal are to 1) investigate the spinal mechanisms for regulation of locomotor circuitry in children with SCI using TcStim, 2) assess whether the combination of task-specific AB-LT and TcStim can acutely potentiate lower limb muscle activity during facilitated stepping, and 3) assess training effects of TcStim combined with AB-LT to promote stepping capacity in non-ambulatory children with SCI.

For this pilot study 8 participants, ages 4-12 years with chronic, acquired SCI, T10 and above and non-ambulatory will be recruited.

For Aim 1, n=8, TcStim will be used to stimulate a single or multi site spinal levels to produce stepping/locomotor activity in lower limbs. Knee, hip, ankle kinematics and electromyography (EMG) of the lower limb muscles in response to stimulation will be recorded during the experiments. The investigators will determine the stimulation parameters that produce rhythmic movements with the greatest increase in lower limb joint excursions as well as EMG amplitude.

For Aim 2, n=8, TcStim will be delivered while participants attempt to take a step overground and while stepping on a computerized treadmill with an overhead partial body weight support (BWS) system. The participants will be stepped at age-appropriate speeds and BWS optimizing the stepping kinematics. The speed and the amount of body weight support provided during the assessment as well as full body kinematics and EMG signals from trunk and lower limb muscles will be recorded during facilitated stepping with and without TcStim.

For Aim 3, n=6, participants will receive 60 sessions of AB-LT+Tcstim. Ability to initiate and complete a step overground with and without stimulation along with full body kinematics and electromyographic (EMG) signals from trunk and lower limb muscles will be recorded at baseline, 20, 40, and 60 sessions of the combined therapy of AB-LT plus TcStim.

ELIGIBILITY:
Inclusion Criteria:

* Children with acquired, upper motor neuron (T10 and above) SCI, traumatic and non-traumatic,
* Chronic injury, defined as greater than one year post injury
* Age 4-12 years,
* Discharged from inpatient rehabilitation,
* Unable to stand, walk, or initiate steps.

Exclusion Criteria:

* Botox use within past 3 months
* Current oral baclofen use,
* Baclofen pump in use,
* Musculoskeletal impairment limiting range of motion, unhealed fracture or other medical complication limiting participation,
* Prior surgery for scoliosis, post SCI
* Congenital SCI,
* Total ventilator dependence.

For Aim 3, additional exclusionary criteria are:

* Unwilling or unable to wean from baclofen during training,
* Use of braces (trunk or lower limb brace).

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Movement observation (live observation) with video review of the ability to initiate and take an independent, voluntary step from a position of standing. | Change in ability to voluntarily step comparing pre-stimulation to during and post stimulation during session 1, session 2, session 3, and session 4 within 1 month of initiation and at session 1, 20, 40, and 60, within a 4 month period
  Ability to take step independently with minimal or no external support. Participant can use a walker or other assistive device for balance and support. The participant will stand independently and lift a limb/foot off the ground and step forward making the same foot contact the ground in front as when taking a first step. This will be measured via movement observation by a licensed physical therapist and videotaped. A single step is all that is required. If more than one step is observed, this information will be documented and also videotaped. No manual assistance will be provided during the assessment for a voluntary step. The achievement of an independent step, foot leaves the ground and is placed forward, is the only criteria for the 'step'.
Electromyography (EMG) recording of lower extremity and trunk muscles | Change in EMG: pre-stimulation compared to during stimulation during session 1, session 2, session 3, and session 4 within 1 month of initiation and at session 1, 20, 40, and 60 within a 4 month period
  Measurement of muscle and nerve functions. The muscle activities are reported in microvolts.
Angular excursions of lower extremity | Change in limb angle excursions: Pre-stimulation compared to during-stimulation during session 1, session 2, session 3, and session 4 within 1 month of initiation and at session 1, 20, 40, and 60 within a 4 month period
  Degrees of flexion/extension, adduction/abduction, and rotation, using wireless motion sensors.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Behrman, PT, PhD, Principal Investigator — University of Louisville
Locations (1):
- Department of Neurosurgery, University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No